CLINICAL TRIAL: NCT02026960
Title: RNA Extraction and Amplification From Biopsy Specimens in Subjects With Metastatic Renal Cell Carcinoma (AGS-NTS-017)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor's clinical program for the agent used in this study was discontinued.
Sponsor: Duke University (Other)
Collaborators: Argos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00047147
Record Dates: First submitted 2014-01-02; First posted 2014-01-03 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Metastatic Renal Cell Carcinoma; Genitourinary Cancer (Bladder, Prostate or Testicular)
MeSH Terms: conditions — Carcinoma, Renal Cell; Urogenital Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal Cell Carcinoma Tumor Tissue (Experimental)
  Interventions: Device: RNA extraction and amplification from biopsy specimens
- Genitourinary tumor tissue (Expansion cohort) (Experimental): Bladder, prostate or testicular cancer
  Interventions: Device: RNA extraction and amplification from biopsy specimens

INTERVENTIONS:
Device: RNA extraction and amplification from biopsy specimens

SUMMARY:
The primary objective is to evaluate methods for AGS-003 production from surgical (stage I) and metastatic biopsy (stage II) Renal Cell Carcinoma (RCC) and a small subset of other GU cancers (expansion cohort) specimens using core needle biopsy in subjects with RCC or other GU cancers. Specifically, this study will evaluate the feasibility of RNA amplification from total tumor RNA isolated from tissues obtained by core needle tumor biopsy.

ELIGIBILITY:
Inclusion Criteria:

A subject with metastatic RCC, who in the opinion of the treating physician, is a potential candidate for inclusion in this study if all of the following criteria apply:

1. 18 years of age or older.
2. Suspected RCC, in the opinion of the investigator
3. Availability of either:

   * Nephrectomy or other surgically removed tissue (Stage I); or,
   * Metastatic RCC biopsy tissue utilizing needle or core biopsy procedures (Stage II).
4. ≥5 biopsy specimens available from BRPC.

   * Subjects who are having a surgical procedure (i.e. metastasectomy, nephrectomy) will have these core biopsies obtained from the surgical specimen, per the BRPC protocol.
5. Not currently being treated with systemic therapy.

Exclusion Criteria:

1. Tumor tissue is committed to other use or inadequate for RNA analysis.
2. Insufficient tissue is collected in the BRPC.

Expansion Cohort for Genitourinary Cancers:

Inclusion Criteria:

1. 18 years of age or older
2. Suspected bladder, prostate, or testicular cancer, in the opinion of the investigator.
3. Availability of surgically removed tissue or biopsy tissue.
4. At least 2 biopsy specimens available from BRPC
5. Not currently being treated with systemic therapy.

Exclusion Criteria:

1. Tumor tissue is committed to other use or inadequate for RNA analysis.
2. Insufficient tissue is collected in the BRPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Success rate for tumor RNA isolation and amplification | At time of surgery or during biopsy
  To Determine the success rate for tumor RNA isolation and amplification create a minimum of 10 doses of AGS-003, as defined by a minimum concentration of ≥84 µg/µL in typically greater than 150 µL final volume RNA. (Tissue obtained at time of surgery or biopsy depending on stage)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harrison, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States